CLINICAL TRIAL: NCT00492479
Title: An Evaluation of Kinerase Pro+Therapy Regimen Vs. Kinerase Vs. Control for the Treatment of Skin Aging
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 5314
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Skin Aging

INTERVENTIONS:
Drug: Kinerase Pro+Therapy Line day repair, serum, night repair
Drug: Kinerase Pro+Therapy Line Ultra rich day repair
Drug: LubriDerm

SUMMARY:
The purpose of this study is to compare the efficacy of the Kinerase Pro+Therapy regimen versus a single Kinerase product vs. control for the treatment of the signs of skin aging.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 35-55 years of age with at least moderate signs of facial aging
* Written informed consent
* Likely to complete all study visits and follow study protocol

Exclusion Criteria:

* Any dermatological or medical condition which would make patient participation unsafe or interfere with study outcomes or measurements
* Known hypersensitivity to any study product or their components
* Recent (within 4 weeks of baseline) surgical treatment to face (including IPL and other laser procedures)
* Prior use of anti-aging treatments for 30 days prior to study entry (physician dispensed or prescribed treatments)
* Planned facial procedures during the study (microdermabrasion, facials, etc)

  o Botox and fillers cannot be used during the trial or for 3 months prior to study entry
* Recent (within 60 days) or concurrent participation in another clinical trial
* Concomitant topical or systemic therapy that my interfere with study measurements or outcomes
* Use of any other topical photoaging/antiaging therapies during the study, other than the prescribed study regimens
* Patients who are habitual tanners (outdoors or with tanning beds) who plan on tanning during the study
* Wearing of cosmetics during study visits

Ages: 35 Years to 55 Years | Sex: Female
Age Groups: Adult
Dates: Start 2007-06; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Yoelin, MD, Principal Investigator — Private Practice
Locations (1):
- Steve Yoelin MD practice, Santa Ana, California, United States